CLINICAL TRIAL: NCT06215248
Title: Assessment of Dysfunction in Left Cardiac Chambers With Strain-analyses in Patients With Lower Extremity Arterial Disease
Brief Title: Myocardial Dysfunction Evaluation in Lower Extremity Arterial Disease Patients With Deformation Analysis
Acronym: MEDAL
Status: Recruiting | Type: Observational
Sponsor: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Jaak Kals, Professor of Vasology, Tartu University Hospital
Other Study IDs: 23105
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Artery Disease; Heart Failure
MeSH Terms: conditions — Peripheral Arterial Disease; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LEAD: LEAD diagnosis confirmed by by ankle-brachial index (≤0,9 or >1,3) or angiography. Fontaine I-IV class symptoms.
- Controls: Matched with LEAD group's patients as much as possible for age, sex, smoking history, hypertension, diabetes, coronary artery disease.

SUMMARY:
Single centre observational study to assess lower extremity arterial disease (LEAD) patients' cardiac dysfunction with strain analyses and to assess connections between cardiac dysfunction, metabolomic changes and target organ damage in LEAD.

ELIGIBILITY:
Inclusion Criteria in LEAD group:

* Fontaine I-IV class symptoms
* Confirmed diagnosis of LEAD

Inclusion Criteria in control group:

* Age 35-85
* Has to have at least of the following: hypertension, diabetes, coronary artery disease or the patient smokes

Exclusion Criteria:

* Age <35 or >85 years
* BMI ≥40 kg/m²
* Known heart failure in history
* Any acute or chronic autoimmune or rheumatic disease
* Cardiac structural disease in history: inflammatory, infiltrative diseases, nonischemic cardiomyopathies
* Acute coronary syndrome in last 3 months
* Moderate to severe cardiac valvular disease
* Cardiac valvular disease operative/invasive treatment in history
* Cardiac implantable electronic device (CIED)
* Transitory ischemic attack or stroke in last 3 months
* Severe COPD (GOLD C or D)
* Moderate to severe asthma (according to GINA 2022 criteria)
* Untreated hypertension (noninvasive blood pressure measurement ≥180/110 mmHg during recruitment)
* Chronic severe kidney dysfunction (eGFR <30 ml/min/1,73 m²)
* Malignant tumor with radiation treatment to thorax, oncologic or biologic treatment in history
* Chronic hematologic disease (except for anemia)
* Severe liver dysfunction
* Malignant tumor with <5 years of remission
* Acute or chronic infectious disease
* Anemia with hemoglobin <80 g/L

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiovascular risk factors
Sampling Method: Non-Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
left ventricular global longitudinal strain (GLS) | after enrollment and one year later
  assessed by deformation analysis with echocardiography

SECONDARY OUTCOMES:
other echocardiographic parameters | after enrollment and one year later
  left ventricular ejection fraction, left atrial strain, lateral, medial and averaged E/E', left atrial volume, maximal tricuspid regurgitation velocity, right ventricular strain
heart failure diagnosis | after enrollment and if necessary, reassessment one year later
  according to European Society of Cardiology year 2021 heart failure guideline (i.e assessment of symptoms, ECG, natriuretic peptides)
arterial stiffness | after enrollment and one year later
  peripheral/central blood pressure, augmentation index, pulse wave velocity in aorta
cardiac- and renal injury markers | after enrollment and one year later
  high-sensitivoty troponin T, natriuretic peptides (NT-proBNP), cystatine C, creatinine, urea, calculated eGFR
metabolomics | after enrollment and one year later
  low molecular weight metabolites
markers of oxidative stress | after enrollment and one year later
  oxidated LDL, interleukine-18, myeloperoxidase, isoprostanes

CONTACTS AND LOCATIONS:
Overall Officials: Jaak Kals, PhD, Principal Investigator — Tartu University Hospital
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Endothelial Research Centre — https://endothelialcentre.ut.ee/